CLINICAL TRIAL: NCT04682990
Title: DIAGNOSIS of PULMONARY TUBERCULOSIS Through HUMAN BREATH TEST Center: Douala - CAMEROON
Brief Title: DIAGNOSIS of PULMONARY TUBERCULOSIS Through HUMAN BREATH (TBENOSE)
Acronym: TBENOSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Yolande Christelle Ketchanji Mougang, Principal Investigator, University of Rome Tor Vergata
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: TB Project eNose-Cameroon
Record Dates: First submitted 2020-12-04; First posted 2020-12-24 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Tuberculosis, Pulmonary; HIV Seropositivity
Keywords: Tuberculosis; Breath test; Volatile Organic Compounds (VOCs)
MeSH Terms: conditions — Tuberculosis, Pulmonary; HIV Seropositivity; Tuberculosis | interventions — Surveys and Questionnaires; Restraint, Physical; X-Rays

STUDY DESIGN:
Intervention Model Description: Positive TB patients (Arm 1) and Negative TB patients (Arm 2 ). All the patients can be HIV positive or not .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary TB (Experimental): This arm will enroll 80-100 patients older than 18 years old, from the Center of Respiratory Diseases in Douala, with pulmonary TB proved by TB LAMP test.
  Interventions:
  1. They will be asked to perform a breath exhalation with a nose clamp.
  2. Medical History: Symptom based Survey, Physical Exam,and HIV status.
  Other interventions:
  * Sputum samples for Ziehl Neelsen smear or Culture in L-J or GeneXpert MTB/RIF;
  * Chest X-ray Follow Up 5 days after beginning of Tx Follow Up 15 days after beginning of Tx Follow Up 30 days after beginning of Tx
  Interventions: Device: Tor Vergata Electronic Nose (TV eNose); Other: Survey & Physical Exam; Diagnostic Test: TB LAMP test; Other: Sputum Samples; Other: Chest X-Ray; Other: Follow Up 5 days after beginning of Tx.; Other: Follow Up & 15 days after beginning of Tx.; Other: Follow Up & 30 days after beginning of Tx.
- Non Pulmonary TB (Active Comparator): This arm will enroll 50-100 patients older than 18 years old, from the Center of Respiratory Diseases in Douala, with Negative pulmonary TB status proved by TB LAMP test. These Negative TB patients can be healthy controls or TB suspects.
  Interventions:
  They will be asked to perform a breath exhalation with a nose clamp. Medical History: Symptom based Survey, and HIV status.
  Other interventions:
  * Sputum samples for Ziehl Neelsen smear or Culture in L-J GeneXpert MTB/RIF;
  * Chest X-ray.
  Interventions: Device: Tor Vergata Electronic Nose (TV eNose); Other: Survey & Physical Exam; Diagnostic Test: TB LAMP test; Other: Sputum Samples; Other: Chest X-Ray

INTERVENTIONS:
Device: Tor Vergata Electronic Nose (TV eNose) — Participants will be asked to perform a breath sampling with a nose clamp in Alveolar sampling bag. This exhaled breath in the sampling bag will be analyse with the TV eNose
Other: Survey & Physical Exam — Perform a oriented survey for risk factors, symptoms and a complete physical exam.
Diagnostic Test: TB LAMP test — Collection of Sputum samples and Perform TB-LAMP (temperature-independent way of amplifying DNA from TB organisms)
Other: Sputum Samples — Sputum samples for Ziehl Neelsen smear or Culture in L-J (if required by the medical staff)
Other: Chest X-Ray — Perform anteroposterior chest X-ray (if required by the medical staff)
Other: Follow Up 5 days after beginning of Tx. — Following the usual planning of the center for Positive TB Patients, they will be asked to come 5 days after initiation of treatment, to perform another measurement with the device.
  Also will perform a Medical History, including Symptom based Survey, Physical Exam, to determine progress of treatment.
  Arms: Pulmonary TB
Other: Follow Up & 15 days after beginning of Tx. — Following the usual planning of the center for Positive TB Patients, they will be asked to come during treatment, to perform another measurement with the device.
  Also will perform a Medical History, including Symptom based Survey, Physical Exam, to determine progress of treatment.
  Arms: Pulmonary TB
Other: Follow Up & 30 days after beginning of Tx. — Following the usual planning of the center for Positive TB Patients, they will be asked to come during treatment, to perform another measurement with the device.
  Also will perform a Medical History, including Symptom based Survey, Physical Exam, to determine progress of treatment.
  Arms: Pulmonary TB

SUMMARY:
Tuberculosis (TB) is one of the top 10 causes of death in the world. More than 95% of TB deaths are in middle- and middle-income countries. Low incomes and long-term diagnosis promote this persistence. In 2017, Cameroon was the 3rd in the top of 20 countries with the highest estimated numbers of incident TB cases among people living with HIV, based on the severity of their TB burden.

World Health Organization (WHO) encourages the introduction of rapid, non-invasive and cheaper screening tests. In this scope, this study proposes the collection of exhaled breath samples and their analysis through the electronic nose made in Tor Vergata University (TV eNose) to diagnose TB and TB-HIV on their participants.

DETAILED DESCRIPTION:
It is a 12 -month dynamic, open, descriptive and analytical type case-control study in adults. The present study intends to recruit , all the Pulmonary TB suspects and case notified by TB Loop-mediated isothermal Amplification(LAMP), sputum culture or GeneXpert Mycobacterium Tuberculosis/Rifampicin (MTB/RIF) Assay, Pulmonary TB+HIV patients, healthy control patients, HIV patients without TB. Each patient will undergo at least two tests: the Breath Test Measurement and the TB LAMP. The TB LAMP will be used like the reference test for positive TB cases.

The enrolment phase of the participants will take 12 months. After this period, additional 6 months will be dedicated to the data analysis and dissemination of results.

Each patient meeting the inclusion criteria will be asked to join the study. Detailed information will be provided him/her. In case of acceptance the participants will undergo further sampling: breath test measurement. All data will be collected ensuring anonymity and privacy. Standard protocols used in the center will not be changed by the research, but each patient will be asked to provide 1 additional sample (exhaled breath in the bag sampler). Each study participant will be properly informed, and a consent form will be signed.

Preparation to participate: It will be required to patients to avoid drinking, eating, smoking, or brushing their teeth 2 hours before the breath test.

Sampling collection: In order to collect breath samples, two bags will be used, one for collecting airways breath (about 0.5 liter volume) and one for alveolar exhaled air (3 liters). It is asked to the patient after putting a clip nose, to inspire with the mouth and to deeply breath inside the bags through an antibacterial filter connected to the sampling apparatus.

At the end, the second bag (volume of 3 liters) contains the alveolar portion of breath that will be analyzed by the TV eNose. During the measurement, the TV eNose will be connected to the computer, to read and store the Volatile Organic Compounds (VOCs) pattern from breath given by the sensor array.

Other data are collected: clinical symptoms, TB LAMP results, and results of others test if available: chest X-ray, smear microscopic, sputum culture and GeneXpert MTB/RIF Assay examinations.

All personal data and results of the patients will be collected in a specific sheet elaborated by the partners (University di Roma Tor Vergata). It will be an Excel database and it will be store in the study site. All data collected will be anonymous.

ELIGIBILITY:
Inclusion Criteria:

* Accept to participate in the study through a signed informed consent approved by the Ethical Committee (CEI of Douala - Cameroon)
* Suspected of having TB on clinical base (4SS + or other clinical suggestions) with HIV+/- status
* Healthy control patient
* Able to produce exhaled air samples
* Able to produce sputum samples for TB LAMP test

Exclusion Criteria:

* Unable to breath normally for 2 minutes due to respiratory illness
* By discretion of the research team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-12-05 (Actual); Study Completion 2021-12-05 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy value of the TV eNose signal value to differentiate patients with Pulmonary TB to control participants | 6 months
  Sensitivity, Specificity and Predictive Values; calculated with an Receiver Operating Characteristic (ROC) curve based on the pattern recognition model from dataset measured by the TV eNose.The classification of the signal is generated with a complex pattern recognition software, using the frequency shift in Hertz (Hz), generated by each of the 12 sensors.
Accuracy value of the diagnostic between Pulmonary TB, Pulmonary TB+ HIV patients and control patients with the TV eNose | 6 months
  Sensitivity, Specificity and Predictive Values; calculated with an Receiver Operating Characteristic (ROC) curve based on the pattern recognition model from dataset measured by the TV eNose. The classification of the signal is generated with a complex pattern recognition software, using the frequency shift in Hertz (Hz), generated by each of the 12 sensors.

SECONDARY OUTCOMES:
Average Days needed to observed a negative result with the device after initiation of treatment. | 6 months
  Get an evolutive model of the VOC pattern of the frequency from each patient under treatment. Characterize VOC pattern of Pulmonary TB with and without treatment

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Palombi, Professor, Study Director — University of Rome Tor Vergata
Locations (1):
- Centre des Maladies Respiratoire, Douala, Littoral Region, Cameroon